CLINICAL TRIAL: NCT05932719
Title: Multicentric Evaluation of COVID-19 Impact on Cancer Patients' Diagnostic and Management: Set-up of Indicators to Follow-up the Activities of Different Cancer Pathologies
Brief Title: Multicentric Evaluation of COVID-19 Impact on Cancer Patients' Diagnostic and Management: Set-up of Indicators
Acronym: COLLAT-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0697
Record Dates: First submitted 2023-07-04; First posted 2023-07-06 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma; Peritoneal Carcinoma
Keywords: COVID-19; Cancer; Health Care Quality Indicators; hepatocellular carcinoma; peritoneal carcinosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peritoneal Carcinosis: Patients hospitalized for peritoneal carcinosis between 2017 and 2020.
  Interventions: Other: COLLAT-COVID is an observational study based on retrospective data issued from patients medial files.
- Hepatocellular Carcinoma: Patients hospitalized for hepatocellular carcinoma between 2017 and 2020.
  Interventions: Other: COLLAT-COVID is an observational study based on retrospective data issued from patients medial files.

INTERVENTIONS:
Other: COLLAT-COVID is an observational study based on retrospective data issued from patients medial files. — The following items will be collected
  * Diagnostic date
  * Diagnostic stage
  * Date of surgery
  * Date of surgery appointment
  * First antineoplastic treatment date
  * Last antineoplastic treatment date
  * Number of treatment cycles recommanded by MDTM

SUMMARY:
The COVID-19 pandemic has deeply and globally impacted usual procedures and patients management in cancer centers. The aim of this study is to set-up and collect indicators to follow-up the activities of different cancer pathologies before and during the pandemic. Patients loss' of chance will be analysed in term of diagnosis and access to care (surgery, antineoplastic treatments).

Data collection will focus on the analysis of 2 specific pathologies for French patients in the "Auvergne-Rhône Alpes" Area: peritoneal carcinosis and hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in France for peritoneal carcinosis or hepatocellular carcinoma between 2017 and 2020.

Exclusion Criteria:

* Patients who did not allow the reuse of their medical data for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in France for peritoneal carcinosis or hepatocellular carcinoma between 2017 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure of patient loss of chance when comparing a set of activity indicators between 2020 and the average activities of previous periods (2017-2019) | 24 months
  The difference between a set of different activity indicators will be compared between 2020 and the average activities of previous periods (2017-2019)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lyon sud, Hospices civils de Lyon, Pierre-Bénite, France